CLINICAL TRIAL: NCT01887782
Title: A Randomized Controlled Study of Conventional Versus Theta Burst Repetitive Transcranial Magnetic Stimulation in the Treatment of Major Depressive Disorder
Brief Title: Randomized Controlled Trial of Conventional vs Theta Burst rTMS
Acronym: HFL vs TBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Daniel Blumberger, Medical Head, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 179/2012
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Major Depressive Disorder
Keywords: depression; magnetic; brain stimulation; treatment-resistant
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HFL rTMS (Experimental): High Frequency Left repetitive transcranial magnetic stimulation five days per week for 4 weeks
  Interventions: Device: HFL rTMS
- iTBS (Active Comparator): intermittent Theta Burst Stimulation (iTBS) five days per week for 4 weeks
  Interventions: Device: iTBS

INTERVENTIONS:
Device: HFL rTMS — Magventure Cool B70 Coil with either RX100 or RX30 Stimulator
  Arms: HFL rTMS
Device: iTBS — Magventure Cool B70 Coil with either RX100 or RX30 Stimulator
  Arms: iTBS

SUMMARY:
This trial will compare a novel form of rTMS, intermittent Theta Burst Stimulation to the standard conventional high frequency left sided stimulation protocol. The Left dorsolateral prefrontal cortex will be the site of stimulation in both treatment conditions. The site of stimulation will be targeted using MRI co-registration. The study seeks to determine if the two treatment protocols have similar effectiveness in treating major depression.

ELIGIBILITY:
Inclusion Criteria:

* outpatients
* voluntary and competent to consent
* Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of MDD, single, recurrent
* between ages 18-65
* failed to achieve a clinical response to an adequate dose of an antidepressant based on an Antidepressant Treatment History Form (ATHF) score of ≥ 3 in the current episode or have been unable to tolerate at least 2 separate trials of antidepressants of inadequate dose and duration (ATHF 1 or 2)
* have a score of ≥ 18 on the HAMD-17 item
* have had no increase or initiation of any psychotropic medication in the 4 weeks prior to screening
* able to adhere to the treatment schedule
* Pass the TMS adult safety screening (TASS) questionnaire
* have normal thyroid functioning based on pre-study blood work

Exclusion Criteria:

* have a history of substance dependence or abuse within the last 3 months
* have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
* have active suicidal intent
* are pregnant
* have a lifetime MINI diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform, delusional disorder, or current psychotic symptoms
* have a MINI diagnosis of obsessive-compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia assessed by a study investigator to be primary and causing greater impairment than MDD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
HAM-D17 score | baseline, after each 5 treatment sessions, and 1, 4, and 12 weeks post-treatment
  Outcome measure is measured by a change in the HAM-D17 score from baseline to week 4 or 6. A 50% improvement in the score is considered response to rTMS. A final score of <8 is categorized as remission.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Blumberger, MD, MSc, Principal Investigator — Centre for Addiction and Mental Health; Jonathan Downar, MD, PhD, Principal Investigator — University Health Network, Toronto Western Hospital; Fidel Vila-Rodriguez, MD, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - Non-Invasive Neurostimulation Therapies Centre, University of British Columbia, Vancouver, British Columbia
  - Toronto Western Hospital, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient level data will be shared once the investigators have completed all proposed analyses from the data set.

REFERENCES:
- [Derived] Kaster TS, Dai Y, Vila-Rodriguez F, Downar J, Daskalakis ZJ, Blumberger DM, Rhee TG. Efficacy of intranasal esketamine versus rTMS for treatment-resistant depression: analysis of individual participant data from two clinical trials. EClinicalMedicine. 2025 Oct 30;90:103609. doi: 10.1016/j.eclinm.2025.103609. eCollection 2025 Dec. PMID 41245530
- [Derived] Kaster TS, Downar J, Vila-Rodriguez F, Baribeau DA, Thorpe KE, Daskalakis ZJ, Blumberger DM. Differential symptom cluster responses to repetitive transcranial magnetic stimulation treatment in depression. EClinicalMedicine. 2022 Dec 2;55:101765. doi: 10.1016/j.eclinm.2022.101765. eCollection 2023 Jan. PMID 36483268
- [Derived] Trevizol AP, Downar J, Vila-Rodriguez F, Thorpe KE, Daskalakis ZJ, Blumberger DM. Predictors of remission after repetitive transcranial magnetic stimulation for the treatment of major depressive disorder: An analysis from the randomised non-inferiority THREE-D trial. EClinicalMedicine. 2020 Apr 30;22:100349. doi: 10.1016/j.eclinm.2020.100349. eCollection 2020 May. PMID 32382720
- [Derived] Ge R, Downar J, Blumberger DM, Daskalakis ZJ, Vila-Rodriguez F. Functional connectivity of the anterior cingulate cortex predicts treatment outcome for rTMS in treatment-resistant depression at 3-month follow-up. Brain Stimul. 2020 Jan-Feb;13(1):206-214. doi: 10.1016/j.brs.2019.10.012. Epub 2019 Oct 18. PMID 31668646
- [Derived] Hsu JH, Downar J, Vila-Rodriguez F, Daskalakis ZJ, Blumberger DM. Impact of prior treatment on remission with intermittent theta burst versus high-frequency repetitive transcranial magnetic stimulation in treatment resistant depression. Brain Stimul. 2019 Nov-Dec;12(6):1553-1555. doi: 10.1016/j.brs.2019.07.011. Epub 2019 Jul 17. PMID 31350213
- [Derived] Kaster TS, Downar J, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Blumberger DM. Trajectories of Response to Dorsolateral Prefrontal rTMS in Major Depression: A THREE-D Study. Am J Psychiatry. 2019 May 1;176(5):367-375. doi: 10.1176/appi.ajp.2018.18091096. Epub 2019 Feb 15. PMID 30764649
- [Derived] Shalbaf R, Brenner C, Pang C, Blumberger DM, Downar J, Daskalakis ZJ, Tham J, Lam RW, Farzan F, Vila-Rodriguez F. Non-linear Entropy Analysis in EEG to Predict Treatment Response to Repetitive Transcranial Magnetic Stimulation in Depression. Front Pharmacol. 2018 Oct 30;9:1188. doi: 10.3389/fphar.2018.01188. eCollection 2018. PMID 30425640
- [Derived] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344